CLINICAL TRIAL: NCT01028807
Title: Early Feeding vs 5-day Fasting After Distal Elective Bowel Anastomoses in Children. A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: ROBERTO DAVILA PEREZ, HOSPITAL INFANTIL DE MEXICO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: robdape2
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2009-12-10 (Estimated); Status verified 2009-12

CONDITIONS: Early Feeding; Bowel Anastomosis
Keywords: Early feeding; Bowel anastomosis; Children

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Experimental group: Early feeding: (Experimental): After 24 hours fasting period, with good abdominal conditions (once flatus passage of bowel movements without abdominal distention, vomiting, nausea or ileus) the oral fluids during 24 hours and then advanced to a regular diet as tolerated.
  Interventions: Other: Early feeding
- Control group : Obligatory 5 day fasting (Active Comparator): Obligatory 5-day fasting because it was the therapeutic gold standard at our hospital and our country. Both groups without NGT and antiemetic drug. 5-day antibiotic regimen, ranitidine and appropriate analgesics were used. Once the regular diet was tolerated, the patients were discharged and followed up at clinic 30 days afterwards.
  Interventions: Other: 5 day fasting

INTERVENTIONS:
Other: Early feeding — after 24 hours fasting period, with good abdominal conditions (once flatus passage of bowel movements without abdominal distention, vomiting, nausea or ileus) the oral fluids during 24 hours and then advanced to a regular diet as tolerated.
  Arms: 1. Experimental group: Early feeding:
Other: 5 day fasting — Obligatory 5-day fasting because it was the therapeutic gold standard at our hospital and our country. Both groups without NGT and antiemetic drug. 5-day antibiotic regimen, ranitidine and appropriate analgesics were used. Once the regular diet was tolerated, the patients were discharged and followed up at clinic 30 days afterwards.
  Arms: Control group : Obligatory 5 day fasting

SUMMARY:
Purpose:

To determine the safety and efficacy of early enteral feeding after distal (ileum-colon) elective bowel anastomoses in children.

Methods:

Controlled randomized trial including all pediatric patients with distal elective bowel anastomosis, excluding non-elective and high risk patients. VARIABLES:

Demographic characteristics, operative time, anastomosis placement,

Follow up: Tolerability variables: beginning peristalsis, beginning bowel movement, time to full diet intake, post-operative stay. Safety variables: mild and persistent vomiting, persistent abdominal distention, wound infection or dehiscence as well as anastomotic leak or dehiscence, reoperation and death. At the end of surgery were randomized to:

1. Experimental group(EG): Early feeding group, after a 24 hours fasting period, with good abdominal conditions (once the post operative ileus had solved), oral fluids and diet was started.
2. Control group (CG): obligatory 5-day fasting. Once the regular diet was tolerated, the patients were discharged. Statistics: Descriptive statistics for global description. Student's t test for quantitative variables and Chi square test for qualitative variables, a p-value less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 1 month to 18 years old that required elective laparotomy with a distal elective bowel anastomosis (ileum and colon).

Exclusion Criteria:

* Proximal and non elective anastomosis
* High risk groups:
* Newborns
* Upper gastrointestinal tract anastomosis (esophagus, gastric, duodenal or jejunal)
* Bilious-digestive or rectal anastomosis
* Immunosuppressed patients
* Gastrostomy or any pre anastomotic derivation
* Multiple anastomoses
* Chronic intestinal obstruction
* Patients who did not complete the minimum POP follow up of one month.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2003-06; Primary Completion 2004-05 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Need to insert a NGT, beginning peristalsis, beginning bowel movement, time to full diet intake, post-operative stay. | First 5 postoperative days

SECONDARY OUTCOMES:
Mild and persistent vomiting, persistent abdominal distention, wound infection or dehiscence as well as anastomotic leak or dehiscence, reoperation and death | First 30 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: ROBERTO DAVILA-PEREZ, SURGEON, Principal Investigator — HOSPITAL INFANTIL DE MEXICO; EDUARDO BRACHO-BLANCHET, SURGEON, Study Chair — HOSPITAL INFANTIL DE MEXICO; JOSE MANUEL TOVILLA-MERCADO, SURGEON, Study Chair — HOSPITAL INFANTIL DE MEXICO; PABLO LEZAMA-DEL-VALLE, SURGEON, Study Chair — HOSPITAL INFANTIL DE MEXICO; GUSTAVO VARELA-FASCINETTO, SURGEON, Study Chair — HOSPITAL INFANTIL DE MEXICO; JAIME NIETO-ZERMEÑO, SURGEON, Study Chair — HOSPITAL INFANTIL DE MEXICO
Locations (1):
- Hospital Infantil de Mexico, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Gokpinar I, Gurleyik E, Pehlivan M, Ozcan O, Ozaydin I, Aslaner A, Demiraran Y, Gultepe M. [Early enteral and glutamine enriched enteral feeding ameliorates healing of colonic anastomosis: experimental study]. Ulus Travma Acil Cerrahi Derg. 2006 Jan;12(1):17-21. Turkish. PMID 16456746
- [Background] Reissman P, Teoh TA, Cohen SM, Weiss EG, Nogueras JJ, Wexner SD. Is early oral feeding safe after elective colorectal surgery? A prospective randomized trial. Ann Surg. 1995 Jul;222(1):73-7. doi: 10.1097/00000658-199507000-00012. PMID 7618972
- [Background] Seenu V, Goel AK. Early oral feeding after elective colorectal surgery: is it safe. Trop Gastroenterol. 1995 Oct-Dec;16(4):72-3. PMID 8854962
- [Background] Senkal M, Mumme A, Eickhoff U, Geier B, Spath G, Wulfert D, Joosten U, Frei A, Kemen M. Early postoperative enteral immunonutrition: clinical outcome and cost-comparison analysis in surgical patients. Crit Care Med. 1997 Sep;25(9):1489-96. doi: 10.1097/00003246-199709000-00015. PMID 9295822
- [Background] Bisgaard T, Kehlet H. Early oral feeding after elective abdominal surgery--what are the issues? Nutrition. 2002 Nov-Dec;18(11-12):944-8. doi: 10.1016/s0899-9007(02)00990-5. PMID 12431715
- [Background] Feo CV, Romanini B, Sortini D, Ragazzi R, Zamboni P, Pansini GC, Liboni A. Early oral feeding after colorectal resection: a randomized controlled study. ANZ J Surg. 2004 May;74(5):298-301. doi: 10.1111/j.1445-1433.2004.02985.x. PMID 15144242
- [Background] Lucha PA Jr, Butler R, Plichta J, Francis M. The economic impact of early enteral feeding in gastrointestinal surgery: a prospective survey of 51 consecutive patients. Am Surg. 2005 Mar;71(3):187-90. PMID 15869128
- [Background] Sangkhathat S, Patrapinyokul S, Tadyathikom K. Early enteral feeding after closure of colostomy in pediatric patients. J Pediatr Surg. 2003 Oct;38(10):1516-9. doi: 10.1016/s0022-3468(03)00506-2. PMID 14577078
- [Background] Pearl ML, Valea FA, Fischer M, Mahler L, Chalas E. A randomized controlled trial of early postoperative feeding in gynecologic oncology patients undergoing intra-abdominal surgery. Obstet Gynecol. 1998 Jul;92(1):94-7. doi: 10.1016/s0029-7844(98)00114-8. PMID 9649101
- [Background] Stewart BT, Woods RJ, Collopy BT, Fink RJ, Mackay JR, Keck JO. Early feeding after elective open colorectal resections: a prospective randomized trial. Aust N Z J Surg. 1998 Feb;68(2):125-8. doi: 10.1111/j.1445-2197.1998.tb04721.x. PMID 9494004
- [Background] Han-Geurts IJ, Hop WC, Kok NF, Lim A, Brouwer KJ, Jeekel J. Randomized clinical trial of the impact of early enteral feeding on postoperative ileus and recovery. Br J Surg. 2007 May;94(5):555-61. doi: 10.1002/bjs.5753. PMID 17443854